CLINICAL TRIAL: NCT04590729
Title: Redistributing Intermittent Physical Activity Breaks to Target Postprandial Glucose Excursion.
Brief Title: Interrupting Sitting Time During Postprandial State
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Franklin Pierce University (Other)
Responsible Party: Principal Investigator, Tongyu Ma, Assistant Professor of Health Sciences, Franklin Pierce University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TM9282020
Record Dates: First submitted 2020-10-11; First posted 2020-10-19 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Sedentary Behavior
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: three-by-three crossover design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3-min Exercise Per 30 Min (Experimental): This protocol involves 3 minutes of cycling on a stationary bike at moderate intensity every 30 minutes for 6 hours, totaling 36 minutes of cycling exercise.
  Interventions: Behavioral: 3-min Exercise Per 30 Min
- 3-min Exercise Per 15 Min (Experimental): This protocol involves 3 minutes of cycling on a stationary bike at moderate intensity every 15 minutes for 3 hours to match the total exercise duration in the first protocol.
  Interventions: Behavioral: 3-min Exercise Per 15 Min
- Sitting (No Intervention): Sitting control.

INTERVENTIONS:
Behavioral: 3-min Exercise Per 30 Min — This protocol involves 3 minutes of cycling on a stationary bike at 50 revolutions per minute and 1 kilopond every 30 minutes for 6 hours, totaling 36 minutes of cycling exercise.
  Arms: 3-min Exercise Per 30 Min
Behavioral: 3-min Exercise Per 15 Min — This protocol involves 3 minutes of cycling on a stationary bike at 50 revolutions per minute and 1 kilopond every 15 minutes for 3 hours, totaling 36 minutes of cycling exercise.
  Arms: 3-min Exercise Per 15 Min

SUMMARY:
The literature has shown that interrupting sitting time with frequent physical activities (e.g., cycling on a stationary bike for 3 minutes every 30 minutes of sitting) is effective for decreasing blood sugar levels. However, the optimal frequency and distribution of sitting interruption remains less clear. The purpose of this study is to compare the effects of two different protocols of sitting interruption (i.e., 3 minutes of cycling every 30 minutes versus 3 minutes of cycling every 15 minutes) on blood sugar levels.

DETAILED DESCRIPTION:
This study will involve two different physical activity conditions and a control condition. Each participant will undergo the three conditions in a random order. The first protocol involves 3 minutes of cycling on a stationary bike at moderate intensity every 30 minutes for 6 hours, totaling 36 minutes of cycling exercise. The second protocol involves 3 minutes of cycling on a stationary bike at moderate intensity every 15 minutes for 3 hours to match the total exercise duration in the first protocol. Participants will remain seated for 3 hours to match to the total time spent in the lab. For the control condition, participants will remain seated. For each condition, participants will be provided with two meals, one before the protocol and another one in the middle of the protocol. The meals will be purchased from the cafeteria on campus based on the participant's own choice as long as carbohydrates account for 55-65% of total calories. Participants will eat identical meals across the three conditions.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy persons
* Sedentary lifestyle

Exclusion Criteria:

* Cardiovascular diseases
* Pulmonary diseases
* Metabolic diseases
* Other contraindications to exercise

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose levels | three and a half hour after the carbohydrates intake
  The investigators will measure capillary blood sugar levels every 30 minutes using the finger-stick method.

CONTACTS AND LOCATIONS:
Overall Officials: Tongyu Ma, Ph.D., Principal Investigator — Franklin Pierce University
Locations (1):
- Franklin Pierce University, Rindge, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No